CLINICAL TRIAL: NCT00001308
Title: Multimodal Studies of Language Production and Comprehension in Normal Volunteers and Patients With Neurologically-Based Language Impairments
Brief Title: Central Mechanisms in Speech Motor Control Studied With H215O PET
Status: Terminated | Type: Observational
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 920178; 92-DC-0178
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2016-10-06

CONDITIONS: Communication Disorder; Healthy; Stuttering; Tourette Syndrome; Voice Disorder
Keywords: Stuttering; Tourette's Syndrome; Spasmodic Dysphonia; Dysarthria; Parkinson's Disease; Verbal Dyspraxia; Aphasia; Speech; Motor Control
MeSH Terms: conditions — Communication Disorders; Stuttering; Tourette Syndrome; Voice Disorders; Dysphonia; Dysarthria; Parkinson Disease; Apraxias; Aphasia; Speech

SUMMARY:
Positron Emission Tomography (PET) is a technique used to investigate the functional activity of the brain. The PET technique allows doctors to study the normal biochemical and metabolic processes of the central nervous system of normal individuals and patients with neurologic illnesses without physical / structural damage to the brain. Radioactive water H215O in PET scans permits good visualization of areas of the brain related to speech.

Most of the PET scan studies conducted have concentrated on learning about how language is formed and decoded. Few studies have been conducted on speech production. This study aims to use radioactive water (H215O) and Positron Emission Tomography (PET scan) to measure blood flow to different areas of the brain in order to better understand the mechanisms involved in speech motor control.

When a region of the brain is active, it uses more fuel in the form of oxygen and sugar (glucose). As the brain uses more fuel it produces more waste products, carbon dioxide and water. Blood carries fuel to the brain and waste products away from the brain. As brain activity increases blood flow to and from the area of activity increases also. Knowing these facts, researchers can use radioactive chemicals (H215O) and PET scans to observe what areas of the brain are receiving more blood flow.

Researchers will ask patients to perform tasks that will affect speech, voice, and language. At the same time patients will undergo a PET scan. The tasks are designed to help researchers observe the blood flow to brain areas associated with voicebox (laryngeal) functions, movement of muscles in the jaw, tongue, and mouth, and other aspects of motor speech.

Special studies will be conducted to evaluate how certain therapies and tasks can draw out symptoms in illnesses in which speech and language are affected. Results of these tests will be used in other studies to evaluate the neurologic mechanisms of diseases like Tourette's syndrome and parkinson's disease.<TAB>

DETAILED DESCRIPTION:
Objective

The primary objective of this protocol is to use multimodal neuroimaging combining complementary electrophysiological and hemodynamic methods to characterize brain-language relationships in healthy subjects and those with neurological disorders that affect speech and language. A secondary objective is to utilize these findings to develop evaluation measures for future treatment studies.

Study Populations

We will focus on four neurological disorders that affect language processing post-stroke aphasia, traumatic brain injury, epilepsy and developmental stuttering. Each constitutes a significant clinical problem central to the NIDCD s mission. These disorders can impair language at several levels - from its elementary perceptual and motor features, the peripheral building blocks of language, to higher levels of language formulation, including word, sentence and narrative processing.

Design

We will utilize a set of tasks designed to evaluate language at the levels at which clinical pathology emerges. We will combine hemodynamic (functional MRI) and electrophysiological (EEG, MEG) modalities to capitalize on the superior spatial resolution of the former and temporal resolution of the latter methods. Whenever possible the same task paradigms are used with both techniques. We will conduct crosssectional sub-studies, addressing specific questions in each of the disorders of interest; we will also conduct longitudinal sub-studies of recovery and neuroplastic reorganization in post-stroke aphasia.

Outcome Measures

Outcome measures include speech-language and psychological tests, measures of behavioral performance during scanning and corresponding MRI, EEG and MEG data. Relationships between these datasets will be evaluated using statistical analytic packages.

ELIGIBILITY:
* INCLUSION CRITERIA FOR ALL SUBJECTS:

Ages 18 to 85.

Ability to provide informed consent.

Must be a Native English speaker by age 2

SPECIFIC INCLUSION CRITERIA FOR SELECTED GROUPS OF HEALTHY VOLUNTEERS:

Have had training and experience in creative writing

Have had training and experience in vocal or instrumental music

Have had training and experience in visual arts

SPECIFIC INCLUSION CRITERIA FOR POST-STROKE APHASIA SUBJECTS:

Had sensorimotor and language deficits following ischemic infarcts.

Had stroke at least two weeks ago.

SPECIFIC INCLUSION CRITERIA FOR TRAUMATIC BRAIN INJURY SUBJECTS:

Diagnosis of TBI

At least one month post-injury

SPECIFIC INCLUSION CRITERIA FOR STUTTERING SUBJECTS:

History of developmental stuttering with symptoms of dysfluency presenting before the age of 13

If recovered, history documented by school or medical records.

SPECIFIC INCLUSION CRITERIA FOR EPILEPSY SUBJECTS:

Ages 18 to 55 years.

Failure of seizures to respond to adequate therapy with at least two standard antiepileptic drugs.

Willingness to be considered for surgery

Fluency in English. Non-native speakers may be included if their fluency is equivalent to that of a native speaker.

Must have localization-related epilepsy

Must be currently enrolled in Protocol 08-N-0161 to participate in this study

EXCLUSION CRITERIA FOR ALL SUBJECTS:

Past or present major medical or psychiatric illnesses (DSM-IV criteria) except Post Traumatic Stress Disorder (PTSD) in TBI subjects an anxiety disorder in stuttering subjects

Significant abnormalities on the general physical examination unrelated to the stroke or TBI

Unable to undergo MRI studies due to pacemakers, aneurysm clips, cochlear implants, shrapnel fragments or a significant history of exposure to small metallic objects which might have become lodged in the tissues of the head or neck or who require hearing aids.

Subjects who are pregnant are excluded from the PET and MRI tests in this study.

Subjects who are lactating are excluded from the PET tests.

Subjects who have or are found to have significant visual agnosia.

Subjects who cannot provide informed consent.

SPECIFIC EXCLUSION CRITERIA FOR POST-STROKE APHASIA SUBJECTS:

More than two prior strokes

Concurrent diagnoses of neurodegenerative disorders or vascular dementia

Comprehension Aphasia Quotient (AQ) of less than 4 on the Western Aphasia Battery (WAB)

SPECIFIC EXCLUSION CRITERIA FOR TRAUMATIC BRAIN INJURY SUBJECTS:

For military subjects: Positive screen for Acinetobacter baumannii-calcoaceticus complex (ABC) infection or colonization

Severe cognitive impairments as evidenced by scores of less than 7 on the Rancho Los Amigos Scale of Cognitive Functioning and/or less than 76 on the Galveston Orientation and Amnesia Test.

For all subjects: Comprehension AQ of less than 4 on the WAB

A diagnosis of PTSD, which is almost always found in TBI subjects recruited from the military, will not disquality TBI subjects from participation.

SPECIFIC EXCLUSION CRITERIA FOR STUTTERING SUBJECTS:

Structural abnormalities on standard clinical (MPRAGE, T2-weighted) MRI scans studies

A diagnosis of anxiety dirorder will not disqualify stuttering subjects from participation

SPECIFIC EXCLUSION CRITERIA FOR EPILEPSY SUBJECTS:

Claustrophobia or anxiety disorders that could be exacerbated by the MRI Scanner

Subjects with neurological disorders, in addition to epilepsy such as, stroke, Parkinson s disease), or who have psychiatric diagnoses (, such as, obsessive-compulsive disorder)

Patients on Phenobarbital or chronic Benxodiazepines

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1163 (Actual)
Dates: Start 1992-04-28; Study Completion 2016-10-06

CONTACTS AND LOCATIONS:
Overall Officials: Allen R Braun, M.D., Principal Investigator — National Institute on Deafness and Other Communication Disorders (NIDCD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Alexander GE, DeLong MR, Strick PL. Parallel organization of functionally segregated circuits linking basal ganglia and cortex. Annu Rev Neurosci. 1986;9:357-81. doi: 10.1146/annurev.ne.09.030186.002041. No abstract available. PMID 3085570
- [Background] Andrews G, Quinn PT, Sorby WA. Stuttering: an investigation into cerebral dominance for speech. J Neurol Neurosurg Psychiatry. 1972 Jun;35(3):414-8. doi: 10.1136/jnnp.35.3.414. PMID 5035315
- [Background] Bartlett EJ, Brown JW, Wolf AP, Brodie JD. Correlations between glucose metabolic rates in brain regions of healthy male adults at rest and during language stimulation. Brain Lang. 1987 Sep;32(1):1-18. doi: 10.1016/0093-934x(87)90115-5. PMID 3498529